CLINICAL TRIAL: NCT07031869
Title: Hand and Wrist Injuries in Professional Hockey Players in Sweden: A Nationwide Observational Cohort Study From the Swedish Hockey League
Brief Title: The Swedish Hockey League Hand and Wrist Injury Tracking Trial
Acronym: SHL-HITT
Status: Active, not recruiting | Type: Observational
Sponsor: Dalarna County Council, Sweden (Other)
Responsible Party: Principal Investigator, Daniel Muder, Principal Investigator, Dalarna County Council, Sweden
Other Study IDs: 2025-01728-01; 2025-01728-01 (Other: Swedish National Ethical Board)
Record Dates: First submitted 2025-06-03; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Register; Injuries; Athletes; Hand Injuries; Wrist Injuries; Prevention
Keywords: hand; wrist; register; athlete; professionel; ice hockey; prevention; SHL; Swedish Hockey League
MeSH Terms: conditions — Wounds and Injuries; Hand Injuries; Wrist Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SHL players with hand/wrist injuries from all games in 2022/23-2024/25 seasons: The study cohort will consist of all registered professional ice hockey players in the Swedish Hockey League (SHL) who have sustained a hand or wrist injury during official SHL games over the course of three full seasons: 2022/23, 2023/24, and 2024/25. This includes players from all 14 teams in the league.
  In total, the study is expected to cover approximately 2,300-2,350 games, including both regular season and playoff matches across the three seasons. All injuries recorded in the SHL's centralized medical injury registry, maintained by the Swedish Medical Association for Ice Hockey, will be included. This registry captures detailed information reported by team medical staff during each season.
  The cohort will include:
  All SHL players active during the 2022/23, 2023/24, and 2024/25 seasons.
  Players of all positions (forwards, defensemen, goalkeepers) and age groups.
  All injuries coded under relevant ICD classifications for trauma to the elbow, forearm, wrist, and han

SUMMARY:
This study, titled Hand and Wrist Injuries in Professional Hockey Players in Sweden: A Nationwide Observational Cohort Study from the Swedish Hockey League (SHL-HITT), aims to deliver a comprehensive national overview of hand and wrist injuries among professional hockey players.

These injuries are relatively common-accounting for approximately 16% of all hockey-related injuries-and can range from minor issues to severe conditions that jeopardize player performance and careers due to prolonged absences or lasting impairment. Despite their significance, there is limited detailed knowledge regarding the specific patterns, mechanisms, and consequences of hand and wrist injuries at the elite level.

Utilizing data from a nationwide injury registry, this observational cohort study will cover three full SHL seasons: 2022/23, 2023/24, and 2024/25. The dataset is expected to include approximately 2,300 games, encompassing both regular season and playoff matches. The study will examine injury characteristics such as type (e.g., fractures, soft tissue damage), player position, in-game timing, and additional contextual factors. Statistical analyses will be conducted to identify trends, correlations, and potential risk profiles among different player groups or positions.

The findings are expected to support the development of enhanced protective equipment and targeted prevention strategies, ultimately contributing to reduced injury incidence and improved athlete health and career sustainability.

The study timeline includes preparation in late 2024, with data collection already ongoing and ethical approval obtained. The analysis will begin following the publication of the study protocol, and we aim for final publication of results in the second half of 2025.

DETAILED DESCRIPTION:
This nationwide observational cohort study, titled Hand and Wrist Injuries in Professional Hockey Players in Sweden: A Nationwide Observational Cohort Study from the Swedish Hockey League (SHL-HITT), aims to systematically characterize the epidemiology and distribution of hand and wrist injuries among elite ice hockey players in the Swedish Hockey League (SHL). Given that upper extremity injuries constitute a significant proportion of hockey-related trauma, with approximately 16% involving the forearm, wrist, and hand, this study addresses a critical gap in the literature regarding the incidence, nature, and severity of these injuries in professional athletes. Utilizing registry data collected since the 2022/23 SHL season, including detailed player baseline characteristics, injury diagnoses classified by ICD codes, and contextual game data, the study will employ descriptive and inferential statistical analyses to elucidate patterns of fracture and soft tissue injuries. Particular emphasis will be placed on evaluating injury mechanisms relative to player position and game situations. Statistical methods will include Pearson correlation, chi-square tests, and parametric or non-parametric tests as appropriate, with significance set at p<0.05. Findings from this study are expected to contribute valuable insights for the development of evidence-based injury prevention strategies and tailored protective interventions aimed at reducing the burden of hand and wrist injuries, thereby potentially enhancing player safety and performance outcomes in professional ice hockey.

ELIGIBILITY:
Inclusion Criteria:

* Professional ice hockey players actively rostered in the Swedish Hockey League (SHL) during the 2022/23 season and onwards.
* Players with recorded forearm, hand or wrist injuries documented in the SHL injury register.

Exclusion Criteria:

* Players not officially signed to an SHL team during the study period.
* Injuries occurring outside the forearm, hand or wrist region.
* Incomplete or missing injury data in the registry.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes professional ice hockey players registered in the Swedish Hockey League (SHL) from the 2022/23 season onward. This cohort encompasses athletes of varying positions who have sustained hand or wrist injuries documented in the league's injury registry.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Distribution and frequency of hand and wrist injuries among professional ice hockey players in the Swedish Hockey League (SHL). | For the 2022/23 to the 2024/25 season.
  Anatomical location (e.g., wrist, hand, fingers, thumb)
  Type of injury (e.g., fracture, dislocation, ligament injury, tendon rupture, contusion)
  Laterality (left vs. right hand)

SECONDARY OUTCOMES:
Injury incidence by player position | For the 2022/23 to the 2024/25 season.
  forward, defenseman, goalie
Time of injury occurrence | For the 2022/23 to the 2024/25 season.
  during game vs. practice; period of the game; season timing
Time lost due to injury | For the 2022/23 to the 2024/25 season.
  number of games missed or duration of absence
Severity of injury | For the 2022/23 to the 2024/25 season.
  The severity of the injuriy will be rated by the time to return to play in days.
  Minimal (1-3 days) Mild (4-7 days) Moderate (8-28 days) Severe (>28 days)
Recurrence of injury | For the 2022/23 to the 2024/25 season.
  Injuries in the same anatomical region during the study period
Baseline characteristics of the cohort | For the 2022/23 to the 2024/25 season.
  Age, stick handedness

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Muder, MD, PhD, Principal Investigator — Center for Clinical Research Dalarna, Uppsala University, Sweden
Locations (1):
- Center for Clinical Research Dalarna, Uppsala University, Sweden, Falun, Dalarna County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Any data shared with colleagues or collaborating researchers will be fully anonymized or pseudonymized to protect participant privacy in accordance with GDPR regulations. Data transfers will occur under strict confidentiality agreements, and all parties will adhere to applicable data protection laws to ensure the security and privacy of personal information. We will act in accordance with the ethical approval granted by the Swedish Ethical Review Authority (EPM) and comply with all relevant local policies regarding data protection.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From the publication of the protocol and for 10 years thereafter.
Access Criteria: Access to individual participant data is typically restricted to authorized researchers involved in the study or approved collaborators under strict confidentiality and data protection agreements.

REFERENCES:
- [Background] Worner T, Kauppinen S, Eek F. Injury patterns in Swedish elite female and male ice hockey - A cross-sectional comparison of past-season's injuries. Phys Ther Sport. 2024 Jan;65:83-89. doi: 10.1016/j.ptsp.2023.12.001. Epub 2023 Dec 8. PMID 38091928
- [Background] Aman M, Forssblad M, Henriksson-Larsen K. Incidence and severity of reported acute sports injuries in 35 sports using insurance registry data. Scand J Med Sci Sports. 2016 Apr;26(4):451-62. doi: 10.1111/sms.12462. Epub 2015 Apr 8. PMID 25850826
- [Background] Toong T, Wilson KE, Urban K, Paniccia M, Hunt AW, Keightley M, Reed N. Grip Strength in Youth Ice Hockey Players: Normative Values and Predictors of Performance. J Strength Cond Res. 2018 Dec;32(12):3494-3502. doi: 10.1519/JSC.0000000000002815. PMID 30216250
- [Background] Jiang R, Westwater ML, Noble S, Rosenblatt M, Dai W, Qi S, Sui J, Calhoun VD, Scheinost D. Associations between grip strength, brain structure, and mental health in > 40,000 participants from the UK Biobank. BMC Med. 2022 Sep 9;20(1):286. doi: 10.1186/s12916-022-02490-2. PMID 36076200
- [Background] Tavares Junior AC, Silva HS, Penedo T, do Amaral Rocha LGS, da Silva AS, Venditti Junior R, Dos-Santos JW. Correlation of the Handgrip Strength and Body Composition Parameters in Young Judokas. Int J Environ Res Public Health. 2023 Feb 2;20(3):2707. doi: 10.3390/ijerph20032707. PMID 36768073